CLINICAL TRIAL: NCT05355922
Title: Efficacy of the Aussie Current Associated With Exercise in the Treatment of Patients With Knee Osteoarthritis: a Randomized, Double-blind Clinical Trial.
Brief Title: Efficacy of the Aussie Current in Patients With Knee Osteoarthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Claudio Cazarini Junior, Doctor of Health Sciences, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Samir Asbahan
Record Dates: First submitted 2021-04-22; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis, Knee; Quadriceps Muscle Atrophy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aussie current (placebo) and Exercises (Sham Comparator)
  Interventions: Other: Electrical electrostimulation of the quadriceps muscle (placebo)
- Aussie current and Exercises (Experimental)
  Interventions: Other: Electrical electrostimulation of the quadriceps muscle

INTERVENTIONS:
Other: Electrical electrostimulation of the quadriceps muscle — Exercises associated with electrical electrostimulation of the quadriceps muscle of patients with knee osteoarthritis
  Arms: Aussie current and Exercises
Other: Electrical electrostimulation of the quadriceps muscle (placebo) — Exercises associated with electrical electrostimulation (placebo) of the quadriceps muscle of patients with knee osteoarthritis
  Arms: Aussie current (placebo) and Exercises

SUMMARY:
Introduction: Osteoarthritis (OA) of the knee is a musculoskeletal disorder and is associated with significant implications related to public health and socioeconomic factors resulting in leave from work. Currently, there are several types of conservative treatment for this pathology, such as medications and mainly muscle strengthening, recommended by international guidelines. It can be associated with neuromuscular electrostimulation (NMES) as with the Aussie Current, for example, which aims to increase strength and function earlier. Objective: To determine whether the effectiveness of adding NMES to the Aussie Current in patients with knee OA who receive treatment based on the principles of conventional physiotherapy, in relation to pain relief, improvement of functional disability and muscle strength. Materials and Method: Forty individuals will be randomly distributed in two groups, with group 1 (G1) exercises and placebo application of electrostimulation and group 2 (G2) exercises and application of NMES with the Aussie current in the quadriceps femoris muscle. In the treatment, 24 sessions will be carried out in a period of 12 weeks based on the gold standard for the treatment of knee OA. Clinical outcomes of pain intensity, functional disability and muscle strength will be measured at baseline, immediately after 12-week treatment and after 24-week follow-up by a single blinded evaluator at all stages. All statistical procedures will be carried out following the principles of "intention to treat" and the comparison between groups will be carried out through the test of Mixed Linear Models. Expected Results: It is expected that there will be improvement in the variables: pain, functional capacity and strength in both the groups, however in the group that carried out the application of the Aussie Current, the gains would be more precocious, when compared to the group that did not carry out the NMES.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of OA in the knees,
* pain for another 06 months
* both genders
* age between 45 and 80 years
* Grade I to III, according to Kellgren-Lawrence.

Exclusion Criteria:

* bearers of severe spine, hip and ankle diseases (fractures and tumors and inflammatory pathologies)
* neurological impairment
* Severe cardiorespiratory diseases

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | Baseline muscle strength (First day)
  Assessment of quadriceps muscle strength with manual dynamometer
Change from Baseline muscle strength at 12 weeks | Change from Baseline muscle strength at 12 weeks
  Assessment of quadriceps muscle strength with manual dynamometer
Change from Baseline muscle strength at 24 weeks | Change from Baseline muscle strength at 24 weeks
  Assessment of quadriceps muscle strength with manual dynamometer
Pain intensity | baseline pain intensity (First day)
  The numerical pain scale
Change from Baseline pain intensity at 12 weeks | Change from Baseline pain intensity at 12 weeks
  The numerical pain scale
Change from Baseline pain intensity at 24 weeks | Change from Baseline pain intensity at 24 weeks
  The numerical pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Cazarini Júnior, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Cittadin GL, Ansolin GZ, Furtado Santana NP, Tonini TL, Buzanello Azevedo MR, de Albuquerque CE, Flor Bertolini GR. Comparison between Russian and Aussie currents in the grip strength and thickness muscles of the non-dominant hand: A double-blind, prospective, randomized-controlled study. Turk J Phys Med Rehabil. 2020 Nov 9;66(4):423-428. doi: 10.5606/tftrd.2020.4718. eCollection 2020 Dec. PMID 33364562
- [Background] Vaz MA, Frasson VB. Low-Frequency Pulsed Current Versus Kilohertz-Frequency Alternating Current: A Scoping Literature Review. Arch Phys Med Rehabil. 2018 Apr;99(4):792-805. doi: 10.1016/j.apmr.2017.12.001. Epub 2017 Dec 14. PMID 29247626